CLINICAL TRIAL: NCT00855972
Title: Low Dose Naltrexone for the Treatment of Juvenile Primary Fibromyalgia Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The FDA IND application is paused due to additional required testing. The IRB protocol was closed prior to research starting.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Principal Investigator, Stanford University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-03022009-1918; 15979
Record Dates: First submitted 2009-03-03; First posted 2009-03-05 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Naltrexone

INTERVENTIONS:
Drug: Low Dose Naltrexone

SUMMARY:
The purpose of this research is to obtain data or information on the safety and effectiveness of low dose naltrexone (LDN) for treating the symptoms of juvenile primary fibromyalgia syndrome. This is a dose finding study to find whether LDN helps the symptoms of juvenile fibromyalgia, and at what dose it does so.

DETAILED DESCRIPTION:
In this pilot dosage-finding and efficacy study, we will experimentally test whether LDN reduces the symptoms of JPFS. We will recruit 40 children with JPFS. Participants will be screened via the JPFS criteria of Yunus and Masi. The study will be an open-label test of various doses of LDN to determine whether LDN reduces JPFS symptoms, and the appropriate dose at which it does so. Primary endpoints will be daily pain, fatigue, and sleep.

The protocol is designed to take 18 weeks. There are a total of 10 study visits, taking place approximately every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:1. Generalized musculoskeletal aching for over 3 months duration 2. Moderate-severe pain in 5 of 11 tender points 3. Age 7 - 17 4. Male or female Exclusion Criteria:1. Diagnosed rheumatic or autoimmune condition contributing to pain 2. Abnormal laboratory results (Rf, ANA, ESR) 3. Use of opioid analgesics in the last 6 months 4. Severe depression and/or anxiety as evidenced by a diagnosis of either disorder, or by evidence based on a clinical interview with the patient and parent at the time of screening. 5. Current or previous psychiatric disorder requiring hospitalization 6. Inability to operate Palm OS® handheld device for self-reports 7. Inability to understand English 8. Inability to attend sessions at Stanford lab every 3 weeks 9. Pregnancy or planned pregnancy, or breastfeeding 10. Abnormal liver functioning tests

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Self Reported Pain | duration of trial
Self-reported fatigue | duration of trial
Overall Fibromyalgia Symptom report | duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Jarred Younger, Sub-Investigator — Stanford University; Sean Mackey, Principal Investigator — Stanford University